CLINICAL TRIAL: NCT06675851
Title: Reward-specific Changes of Cerebral Dopamine Synthesis in Healthy Volunteers and Depressed Patients
Brief Title: Reward-specific Changes of the Chemical Messenger Dopamine in the Brain of Healthy and Depressed People
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Austrian Science Fund (FWF) (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, Univ.-Prof. Priv.-Doz. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2321/2019; 2019-004880-33 (EudraCT Number)
Record Dates: First submitted 2024-10-31; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: functional PET; PET/MRI; Reward; Bupropion; Escitalopram; MDD; Depression; nucleus accumbens; dopamine synthesis; FDOPA
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Bupropion; halofantrine; Dexetimide; Escitalopram

STUDY DESIGN:
Intervention Model Description: Double-blind, prospective, longitudinal (optional cross-over-design in selected patients)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Antidepressant treatment in MDD patients with bupropion (Active Comparator): Bupropion 150 mg daily after baseline PET/MRI or MRI/MRS over 6-8 weeks
  Interventions: Drug: WELLBUTRIN SR (Bupropion HCI) Sustained-Release Tablets, 150 mg; GlaxoSmithKline
- Antidepressant treatment in MDD patients with escitalopram (Active Comparator): Escitalopram 10 mg daily after baseline PET/MRI or MRI/MRS over 6-8 weeks
  Interventions: Drug: Cipralex (escitalopram)
- Healthy Controls without antidepressant intake (No Intervention): Healthy controls will only attend imaging procedures without medication intake

INTERVENTIONS:
Drug: WELLBUTRIN SR (Bupropion HCI) Sustained-Release Tablets, 150 mg; GlaxoSmithKline — Bupropion 150 mg daily after baseline PET/MRI or MRI/MRS over 6-8 weeks
  Arms: Antidepressant treatment in MDD patients with bupropion
Drug: Cipralex (escitalopram) — Escitalopram 10 mg daily after baseline PET/MRI or MRI/MRS over 6-8 weeks
  Arms: Antidepressant treatment in MDD patients with escitalopram

SUMMARY:
Major depressive disorder was shown to be associated with pathological alterations within neurotransmitter systems of the brain. Based on earlier study results, it is assumed that the neurotransmitter dopamine is relevant for several symptoms of depression, e.g., loss of interest or pleasure and lack of motivation. Thus, it is assumed that the synthesis of dopamine in the brain of depressed individuals could be impaired. The specific effect of common antidepressants on the human reward system in depression has not yet been sufficiently investigated. In particular, it is unclear whether depressed patients exhibit reward-specific changes of dopamine synthesis, and whether or not these changes can be differentially affected by diverse types of antidepressants. Neurotransmitter systems can be visualized in the brain using positron emission tomography (PET). Additionally, brain structure and function can be studied using magnetic resonance imaging (MRI). For the visualization of dopamine synthesis in the brain, the radioligand [18F]FDOPA can be used in PET measurements. To assess task-relevant changes of diverse radioligands and thus specific metabolic processes in the brain during specific tasks, a recently developed PET-approach can be used which has already been successfully applied in a pilot study with healthy volunteers. In the present project, 60 depressed subjects and 30 healthy controls will undergo PET/MR-imaging twice. Depressed subjects will be assigned to 1 of 2 treatment groups. 30 depressive subjects will receive bupropion, the other 30 patients will be treated with escitalopram. After a treatment period of 6 weeks, the 2nd PET measurement will be performed in all participants, aiming to detect potential reward-specific changes of dopamine synthesis. The investigators hypothesize that reward-specific changes of dopamine synthesis will be lower in depressed subjects than in healthy controls, that reward-specific changes of dopamine synthesis will be significantly higher in the bupropion group than in the escitalopram group, and that the changes of dopamine synthesis will be associated with functional changes in the brain (measured by simultaneous functional MRI scans). This will be the first study comparing the effects of escitalopram and bupropion on task-specific dopamine synthesis and thus on the human reward system. The study is expected to yield new insights for individual treatment concepts in the therapy of depression.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged between 18-65 years of age
* Depressive patients: DSM-IV diagnosis of MDD following SCID I, HDRS29, MADRS and BDI-II
* Satisfactory general health as determined by past medical history, physical examination, vital signs at screening
* Vital signs measured after 3 minutes resting in the supine position must be within the following ranges: oral body temperature between 35.0-37.5 °C, systolic blood pressure 90-140 mmHg, diastolic blood pressure 50-90 mm Hg, pulse rate 40-100 bpm
* Subjects must weigh 50-100 kg to participate in this study with a BMI within 19-26.
* Sufficient visual and auditory performance for neuropsychological testing
* Written informed consent will be obtained prior to the start of any study procedures. Therefore, willingness and competence to sign the informed consent form is needed.
* Potential patients must be able to communicate well with the investigator and comply with the requirements of the study
* Only participants who are legally authorized to give informed consent will be included in the present study.

Exclusion Criteria:

* Depressed patients: Presence of any severe / unstable neurological, somatic or psychiatric comorbidity
* Healthy controls: Any psychiatric disease or any severe / unstable neurological or somatic disease
* Presence of psychotic symptoms
* Acute suicidality
* Any contraindication for magnetic resonance or PET imaging
* Presence of any metallic implant in the head
* History of clinically significant drug allergy; history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to one of the study drugs or multiple study drugs (known hypersensitivity to bupropion, escitalopram)
* Other clinically significant abnormality on physical, neurological, or laboratory examination or on electrocardiogram (ECG) that, in the opinion of the investigator precludes the patient from the study
* Ingestion of antidepressants or other psychotropic agents within the last 6 months Previous escitalopram- or bupropion intake
* Antidepressive trials wit DBS, electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS) or Ketamine
* Current smoking, substance abuse including alcohol, drugs of abuse, or any medication in a manner which is indicative of substance-related disorders (e.g. substance dependency) according to DSM-IV
* Failure to comply with the study protocol or follow the instructions of the investigators
* Positive urine pregnancy test
* Known pregnancy or lactation
* MRI scan that shows evidence of stroke, infarct, or other space occupying lesion or structural abnormality
* History of any other drug or alcohol abuse or misuse
* Participation in any clinical investigation within 12 weeks prior to dosing
* Evidence from an Allen test of incomplete communication between the radial and ulnar artery, in either hand
* Significant radiation exposure (>5 mSv) in the frame of participation in trials within the past 10 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes of the reward specific dopamine synthesis rate in the nucleus accumbens of depressed individuals after 6-8 weeks of antidepressant intake assessed via functional PET | 6-8 weeks
  Reward-specific dopamine synthesis rate: Assessment of the net influx constant Ki in the nucleus accumbens via functional PET using [18F]FDOPA as an index of the dopamine synthesis rate
Relationship between potential changes of the reward-specific dopamine synthesis rate in the nucleus accumbens assessed via functional PET and treatment response in depressed individuals after 6-8 weeks of antidepressant intake | 6-8 weeks
  Reward-specific dopamine synthesis rate: Assessment of the net influx constant Ki in the nucleus accumbens via functional PET using [18F]FDOPA as an index of the dopamine synthesis rate; Treatment response rates will be assessed at baseline and after 6-8 weeks of antidepressant therapy via the Hamilton Depression Rating Scale with 29 items (HDRS29) and the Montgomery-Åsberg Depression Rating Scale (MADRS).
Difference in changes to the reward-specific dopamine synthesis rate in the nucleus accumbens assessed via functional PET in depressed patients taking bupropion vs. escitalopram after 6-8 weeks of therapy | 6-8 weeks
  Reward-specific dopamine synthesis rate: Assessment of the net influx constant Ki in the nucleus accumbens via functional PET using [18F]FDOPA as an index of the dopamine synthesis rate

SECONDARY OUTCOMES:
Relationship between the reward-specific dopamine synthesis rate (assessed via functional PET) and fMRI activation across healthy volunteers and depressed patients, both at baseline and after 6-8 weeks of therapy | 6-8 weeks
  Reward-specific dopamine synthesis rate: Assessment of the net influx constant Ki in the nucleus accumbens via functional PET using [18F]FDOPA as an index of the dopamine synthesis rate; fMRI activation: Blood-Oxygenation-Level Dependent Signal via functional Magnetic Resonance Imaging
Remission rates in depressed patients being treated with either escitalopram or bupropion in a longitudinal design | 6-8 weeks
  Remission rates will be assessed at baseline and after 6-8 weeks of antidepressant therapy via the Hamilton Depression Rating Scale with 29 items (HDRS29) and the Montgomery-Åsberg Depression Rating Scale (MADRS).
Test-retest reliability for the quantification of dopamine synthesis rates in healthy volunteers via functional PET | 6-8 weeks
  Reward-specific dopamine synthesis rate: Assessment of the net influx constant Ki in the nucleus accumbens via functional PET using [18F]FDOPA as an index of the dopamine synthesis rate; assessed at baseline and after 6-8 weeks without any interventions in between

OTHER OUTCOMES:
Changes in cerebral GABA and Glutamate after antidepressant treatment measured by Magnetic Resonance Spectroscopy (MRS) | 6-8 weeks
  GABA+/tCr, GABA+/Glx, and Glx/tCr ratios will be assessed via MRS before and after antidepressant treatment over 6-8 weeks. This will be an optional measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reed MB, Handschuh PA, Schmidt C, Murgas M, Gomola D, Milz C, Klug S, Eggerstorfer B, Aichinger L, Godbersen GM, Nics L, Traub-Weidinger T, Hacker M, Lanzenberger R, Hahn A. Validation of cardiac image-derived input functions for functional PET quantification. Eur J Nucl Med Mol Imaging. 2024 Jul;51(9):2625-2637. doi: 10.1007/s00259-024-06716-8. Epub 2024 Apr 27. PMID 38676734
- See also: Related Info — https://www.fwf.ac.at/forschungsradar/10.55776/KLI1006